CLINICAL TRIAL: NCT03455075
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind Trial of Spermatogenesis Suppression After Oral Administration of Dimethandrolone Undecanote (DMAU) Alone or With Levonorgestrel (LNG) for 12 Weeks Versus Placebo Alone in Normal Men
Brief Title: Study of Spermatogenesis Suppression With DMAU Alone or With LNG Versus Placebo Alone in Normal Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CCN010B
Record Dates: First submitted 2018-02-22; First posted 2018-03-06 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Healthy; Men; Male Contraception
Keywords: Healthy Men; Male Contraception; Androgen; Dimethandrolone; Levonorgestrel
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — dimethandrolone-undecanoate; Levonorgestrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Lower DMAU + LNG (Experimental): DMAU 100 mg + LNG 30 mcg administered orally in capsules.
  Interventions: Drug: Dimethandrolone-Undecanoate; Drug: Levonorgestrel 0.03 MG
- Middle DMAU + LNG (Experimental): DMAU 200 mg + LNG 30 mcg administered orally in capsules.
  Interventions: Drug: Dimethandrolone-Undecanoate; Drug: Levonorgestrel 0.03 MG
- Middle DMAU + Placebo (Experimental): DMAU 200 mg + placebo administered orally in capsules.
  Interventions: Drug: Dimethandrolone-Undecanoate; Drug: Placebo oral capsule
- Higher DMAU + Placebo (Experimental): DMAU 400 mg + placebo administered orally in capsules.
  Interventions: Drug: Dimethandrolone-Undecanoate; Drug: Placebo oral capsule
- Placebo (Placebo Comparator): Placebo administered orally capsules.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Dimethandrolone-Undecanoate — Single doses of DMAU in castor oil/benzyl benzoate administered in 100 mg capsules.
  Other Names: DMAU
  Arms: Higher DMAU + Placebo; Lower DMAU + LNG; Middle DMAU + LNG; Middle DMAU + Placebo
Drug: Levonorgestrel 0.03 MG — Single doses of LNG administered in 30 mcg capsules.
  Other Names: LNG
  Arms: Lower DMAU + LNG; Middle DMAU + LNG
Drug: Placebo oral capsule — Placebo capsules that look like DMAU and LNG capsules but with no active ingredients.
  Arms: Higher DMAU + Placebo; Middle DMAU + Placebo; Placebo

SUMMARY:
This is a Phase IIa multicenter, double-blind, placebo-controlled study in healthy men to evaluate the spermatogenesis suppression after oral administration of Dimethandrolone Undecanoate (DMAU) alone or with Levonorgestrel (LNG) for 12 weeks versus placebo alone.

DETAILED DESCRIPTION:
This 12 week repeated dose study will be conducted at two centers: the Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center and the University of Washington. The sites propose to enroll approximately 100 men with a goal of enrolling 20 healthy male subjects in each of the 4 active groups and 20 in the placebo group for 12 weeks of treatment. The goal is to complete at least 17 efficacy evaluable subjects in each group. The DMAU for this study will be castor oil formulation administered after a 25 to 30 g fat meal. The oral dose of LNG will be 30 mcg per day. The study volunteers will be randomized to one of five treatment groups:

Group 1: Lower DMAU dose (100 mg per day) + LNG (30 mcg per day) (n=20) Group 2: Middle DMAU dose (200mg per day) + LNG (30 mcg per day) (n=20) Group 3: Middle DMAU dose (200 mg per day) + placebo LNG (n=20) Group 4: Higher DMAU dose (400 mg per day) + placebo LNG (n=20) Group 5: Placebo DMAU capsules and placebo LNG capsules (n=20)

Each treatment group will receive the identical number of capsules in blinded fashion so that each subject will receive an identical number of capsules in order to maintain the blind.

ELIGIBILITY:
Men who meet all the following criteria are eligible for enrollment in the trial:

1. Male volunteers in good health as confirmed by physical examination, medical history, and clinical laboratory tests of blood and urine at the time of screening.
2. 18 to 50 years of age (inclusive) at the time of the screening visit.
3. BMI ≤36 calculated as weight in kg/ (height in m2).
4. No history of steroid hormone use in the three months prior to the first screening visit or any current medication use which might interfere with steroid metabolism.
5. Subject agrees to use a recognized effective method of contraception with any female partner (refer to Appendix 7 for acceptable forms of contraception) during the course of the study treatment and recovery phases until recovery is confirmed and study exit occurs.
6. Subjects will refrain from donating blood or plasma during the study period and from participating in other investigational drug studies.
7. Subjects will be advised to refrain from excessive alcoholic consumption during the study period. (No more than 15 drinks per week and no alcohol consumption within 24 hours of a study visit.)
8. Subjects will be advised to refrain from excessive marijuana consumption during the study period. (No more than 3 uses per week and no consumption within 24 hours of a study visit.)
9. No known or suspected current alcohol dependence syndrome, chronic marijuana use, or any illicit drug use that may affect metabolism/transformation of steroid hormones and study treatment compliance.
10. Subjects will be advised to refrain/abstain from grapefruit juice during the study period.
11. In the opinion of the investigator, subject is able to comply with the protocol, understand and sign an informed consent and HIPAA form.
12. Subjects will be advised to refrain from major changes in their level of exercise during the study period.

Men who meet any of the following criteria are NOT eligible for enrollment in the trial:

1. Men participating in another clinical trial involving an investigational drug within the 30 days prior to the first screening visit.
2. Men not living in the catchment area of the clinic or within a reasonable distance from the study site.
3. Clinically significant abnormal physical or laboratory findings at screening.
4. Elevated PSA (levels ≥ 2.5 ng/mL) at screening, according to local laboratory normal values.
5. IPSS score ≥ 10.
6. Abnormal serum chemistry values at screening, according to local laboratory reference ranges that indicate liver or kidney dysfunction or that may be considered clinically significant. In addition, the following upper limits will be observed: fasting bilirubin less than 2 mg/dL, cholesterol less than 221 mg/dL, and fasting triglycerides less than 201 mg/dL.
7. Abnormal semen analyses or abnormal semen concentration as defined by the WHO semen manual (< 15 million/mL).
8. Use of androgens within 3 months before first screening visit except for long acting testosterone which requires a wash out period of 4 months prior to screening.
9. Ongoing use of androgens or other compounds for body building including nutritional supplements.
10. Systolic BP ≥130 mm Hg and Diastolic blood pressure BP ≥ 80 and mm Hg; Blood pressure (BP) will be taken 3 times at 5 - minute intervals and the mean of second and third measurements will be used to determine eligibility. (Note: Diagnosis of hypertension or treatment of hypertension is exclusionary.)
11. PHQ-9 score of 15 or above.
12. History of hypertension, including hypertension controlled with treatment.
13. Known history of primary testicular disease or disorders of the hypothalamic-pituitary axis.
14. Benign or malignant liver tumors; active liver disease.
15. History of breast carcinoma.
16. Known history of androgen deficiency due to hypothalamic-pituitary or testicular disease.
17. Known history of cardiovascular, renal, hepatic or prostatic disease or significant psychiatric illness.
18. Positive serology for active Hepatitis (not immunization-related serology) or HIV at screening visit.
19. A serious systemic disease such as diabetes mellitus.
20. History of known, untreated sleep apnea.
21. Partner is known to be pregnant.
22. Men desiring fertility within 12 months of signing consent for study participation.
23. Men participating in competitive sports where drug screening for prohibited substances (including anabolic steroids) is routine. Exclusion is due to the potential of testing positive for androgens that may occur from their study participation coupled with the unknown efficacy (i.e. duration of positive testing) from 12-week daily use of DMAU.
24. Use of sex steroids or medications which might interfere with steroid metabolism (i.e. ketoconazole, finasteride, oral corticosteroids, dutasteride and statins).
25. Use of medications that will interfere or interact with DMAU or LNG.
26. Known hypersensitivity to any of the active substances of DMAU, of the excipients of the study treatment, or LNG.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 92 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Suppression of spermatogenesis as assessed by semen analyses using number of subjects with sperm concentration <3 million (M)/mL with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks

SECONDARY OUTCOMES:
Assessing suppression of gonadotropins using percentage of subjects with FSH and LH ≤ 1.0 IU/L. | 2 months
Changes from baseline in sperm concentration. | 4 - 6 months
Changes from baseline in LH level. | 4 - 6 months
Changes from baseline in FSH level. | 4 - 6 months
Changes from baseline in Testosterone level. | 4 - 6 months
Changes from baseline in Estradiol level. | 4 - 6 months
Changes from baseline in DHT level. | 4 - 6 months
Changes from baseline in SHBG level. | 4 - 6 months
Changes from baseline in DMA level. | 4 - 6 months
Changes from baseline in DMAU level. | 4 - 6 months
Changes from baseline in LNG level. | 4 - 6 months
Incidence of treatment emergent adverse events (safety and tolerability) with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in sodium with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in potassium with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in bicarbonate with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in chloride with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in fasting glucose with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in blood urea nitrogen with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in creatinine with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in calcium with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in total bilirubin with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in alkaline phosphatase with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in alanine aminotransferase with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in aspartate transaminase with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in albumin with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in PSA with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone. | 12 weeks
Changes from baseline in sexual function with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone using the psychosexual daily questionnaire. | 12 weeks
Changes from baseline in prostate function with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone using the International Prostate Symptom Score. | 12 weeks
Changes from baseline in mood with daily oral dose of DMAU (3 different doses) alone or with LNG 30 mcg for 12 weeks versus placebo alone using the Patient Health Questionnaire-9. | 12 weeks
Changes from baseline in blood pressure. | 4 - 6 months
Changes from baseline in heart rate. | 4 - 6 months
Changes from baseline in weight. | 4 - 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Washington Medical Center & Health Sciences, Seattle, Washington